CLINICAL TRIAL: NCT07315074
Title: Effect of Esketamine on Postoperative Sleep in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, MD, the Deputy Director of Anesthesiology, the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20251115
Record Dates: First submitted 2025-12-04; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Circadian Rhythm; Postoperative Sleep Disturbance
Keywords: Esketamine; Circadian Rhythm; Melatonin; Postoperative Sleep Disturbance; Postmenopause
MeSH Terms: interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine Group (Group E) (Experimental)
  Interventions: Drug: Esketamine
- Control Group (Group C) (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Esketamine — Participants in Group E are administered esketamine with a loading dose of 0.2 mg/kg (diluted to 10 ml with normal saline) and a maintenance dose of 0.2 mg·kg-¹·h-¹ .
  Arms: Esketamine Group (Group E)
Drug: Normal Saline — In Group C, a loading dose of normal saline 10 ml and a maintenance dose of 10 ml/h of normal saline is given intravenously.
  Arms: Control Group (Group C)

SUMMARY:
The prevalence of sleep disturbance among postmenopausal women has been reported to reach 51.6%. Epidemiological studies consistently show that the incidence of sleep disorders increases with age and menopausal transition. Compared with premenopausal women, postmenopausal women demonstrate reduced circadian rhythm stability and a higher prevalence of sleep disturbance. In this population, levels of melatonin, total sleep time, sleep latency, N3 stage sleep, and the circadian amplitude of alertness are all diminished. Sleep disturbance can adversely affect both the mental and physical health of women and significantly impair their social functioning. Poor sleep is associated with decreased cognitive performance and heightened emotional distress, contributing to diminished quality of life. Moreover, prolonged sleep deprivation elevates the risk of developing obesity, diabetes, cardiovascular conditions, and psychiatric disorders.

Circadian rhythms are endogenous physiological and behavioral cycles that oscillate over approximately 24 hours, governing critical processes such as sleep-wake cycles, hormonal fluctuations (e.g., cortisol and melatonin). These rhythms are regulated by the suprachiasmatic nucleus (SCN). Disruptions in circadian rhythms have been associated with sleep disturbances.

Esketamine is the S (+) enantiomer of ketamine and has a higher affinity for the NMDA receptor than the R-enantiomer. Previous studies have demonstrated that intraoperative administration of esketamine can improve postoperative sleep quality and reduce the incidence of postoperative sleep disturbances, through its antidepressant efficacy, anti-inflammatory properties, analgesic efficacy, neurocognitive and anxiolytic effects. However, few studies have investigated whether esketamine can regulate circadian rhythms and subsequently affect sleep, especially in postmenopausal women.

The objective of this two-center, prospective, randomized controlled clinical trial is to investigate the effects of esketamine on postoperative sleep in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I-III.
2. Postmenopausal women (aged > 40 years, postmenopause for more than 12 months; excluding pregnancy).
3. Aged > 40 years.
4. Scheduled to undergo elective lower-limb fracture surgery under general anesthesia.
5. Body Mass Index (BMI) between 18 and 28 kg/m².
6. Expected surgical duration of ≥ 60 min.
7. Patients who require perioperative urinary catheterization.

Exclusion Criteria:

1. Presence of preoperative sleep-related disorders, such as obstructive sleep apnea or restless legs syndrome.
2. History of drug or alcohol abuse or dependence.
3. Known contraindications or allergies to esketamine or other anesthetic agents.
4. Use of psychotropic medications or sex hormones within the past 3 months.
5. Shift work or taking medications affecting melatonin.
6. Severe comorbid conditions, including but not limited to: uncontrolled hypertension, coronary artery disease, cardiac insufficiency, pulmonary hypertension, intracranial hypertension or elevated intraocular pressure, hyperthyroidism, severe hepatic or renal dysfunction.
7. History of cerebral infarction, intracerebral hemorrhage, or residual central nervous system deficits.
8. History of uterine or ovarian surgery.
9. Impairments of language, hearing, vision, or cognitive function that would prevent completion of questionnaires or cooperation with sleep monitoring.
10. Transfer to ICU postoperatively.

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative sleep disturbance | Postoperative day 1.
  The primary outcome is the incidence of postoperative sleep disturbance (PSD) , evaluated using the Numeric Rating Scale (NRS) and the Athens Insomnia Scale (AIS) on postoperative day 1. PSD is defined as an NRS score of 6 or higher or an AIS score of 6 or higher.

SECONDARY OUTCOMES:
Biological rhythm detection | From preoperative day 1 to postoperative day 3.
  Melatonin rhythm profiles are analyzed using saliva samples by measuring melatonin every 6 h for 48 h: at 10:00 PM on the night of surgery; 4:00 AM, 10:00 AM, 4:00 PM, and 10:00 PM on postoperative day 1; and 4:00 AM and 10:00 AM on postoperative day 2.
  Expression of core circadian clock genes (CLOCK, BMAL1, PER1, PER2, CRY1, CRY2) and blood melatonin concentrations are assessed on preoperative day 1, postoperative day 1 and postoperative day 3.
PSQI | Preoperative day 1 and postoperative day 30.
  Subjective sleep quality, sleep length, sleep latency, habitual sleep efficiency, use of sleep drugs, sleep disruptions, and daytime dysfunction are among the seven domains in which the 19 items are assessed. A scale of 0 to 3 is utilized to grade the domains, with 3 denoting serious impairment. The seven subscale scores are then added together to generate a global PSQI score, which ranged from 0 to 21 points, with a total score greater than 7 indicates poor sleep quality.
Objective sleep parameters recorded by actigraphy | From preoperative day 1 to postoperative day 3.
  Objective sleep parameters will be recorded using actigraphy.The parameters include total sleep time (TST), sleep onset latency (SOL), wake after sleep onset (WASO), proportion of WASO (WASO%), and sleep efficiency (SE%).
Anxiety and Depression assessments | From preoperative day 1 to postoperative day 30.
  Anxiety and depression are measured using the Hospital Anxiety and Depression Scale (HADS). It comprises two subscales: the Anxiety subscale (HADS-A) and the Depression subscale (HADS-D). For each item, respondents select the degree of severity, ranging from 0 to 3, representing none, mild, moderate, and severe. The total score for each subscale ranges from 0 to 21, with higher scores indicating more severe anxiety or depression symptoms. Scores of 0-7 are considered normal, 8-10 suggest the possibility of mild anxiety or depression, 11-14 indicate the possibility of moderate anxiety or depression, and 15-21 signify the possibility of severe anxiety or depression.
Frontal electroencephalography | From entering the operating room to surgery ending.
  Electroencephalogram (EEG) data is collected using the ConView Anesthesia Depth Monitoring System (ConView YY-105, Zhejiang Puke Medical Technology Co., Ltd., China). The analysis includes the power spectrum of EEG energy across various frequency bands, the peak frequencies in the α-β band, and key electrocorticogram indices such as the left α-index (Aileft), right α-index (Airight), electromyographic index (EMG), and burst suppression ratio (BSR).
Postoperative cognitive function and biomarkers | From preoperative day 1 to postoperative day 3.
  Delirium assessments is conducted twice daily on postoperative days 1, 2, and 3 with at least 6 hours between evaluations, using the Chinese version of the 3-Minute Diagnostic Confusion Assessment Method (3D-CAM).
  Brain-derived neurotrophic factor (BDNF) and S100β are measured from blood samples collected on preoperative day 1, postoperative day 1 and postoperative day 3.
Inflammatory markers | From preoperative day 1 to postoperative day 3.
  Inflammatory biomarkers including tumor necrosis factor-α (TNF-α), interleukin (IL)-1β, IL-6, and IL-10 are measured.
Postoperative pain assessment | From postoperative day 1 to day 3.
  Pain levels, including both rest and exercise pain, are measured using the Visual Analogue Scale (VAS) at 24 hours, 48 hours, and 72 hours postoperatively. Data on the use of the Patient-Controlled Analgesia (PCIA) device, including trigger times for bolus doses within the first 24 hours post-surgery the total number of bolus presses, and the use of the rescue analgesic flurbiprofen, are documented.

OTHER OUTCOMES:
Possible adverse reactions | From esketamine infusion to postoperative day 3.
Heamodynamics | From entering the operating room to surgery ending.
  Heart rate (HR) is recorded at the following time points: 5 minutes after patient entry, during intubation, at the start of surgery, and at the end of surgery.
Heamodynamics - mean arterial pressure (MAP) | From entering the operating room to surgery ending.
  Mean arterial pressure (MAP) is recorded at the following time points: 5 minutes after patient entry, during intubation, at the start of surgery, and at the end of surgery.
Quality of postoperative recovery | From postoperative day 1 to day 3.
  The QoR-15 score is used to assess the quality of recovery. The QoR-15 includes five dimensions: physical comfort, physical independence, emotional state, pain, and psychological support, with a total of 15 questions. Each question is scored from 0 to 10, with a higher score indicating better recovery quality.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jingjiang People's Hospital, Jingjiang, Jiangsu
  - The Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No